CLINICAL TRIAL: NCT04016584
Title: Diabetes Pueblo Program - The Application and Acceptability of Culturally Appropriate Education Programs for Current or Potential Insulin Therapy Users With Type 2 Diabetes in the Latino Community
Brief Title: Diabetes Pueblo Program - Application and Acceptability of Culturally Appropriate Latino Education for Insulin Therapy
Acronym: DiabPueblo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY2017-6000
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Type2 Diabetes
Keywords: Type 2 Diabetes; Latino/Hispanic; Promotore; Community health worker
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Latino adults with type 2 diabetes (Experimental): Participants of the Diabetes Pueblo Education Program will include adults with T2D from the Santa Barbara Latino community whose diabetes is poorly controlled, defined as -
  1. hemoglobin A1c > 8% at or prior to enrollment, or
  2. hemoglobin A1c < 8% (within the last 3 months), AND with at least one of the following (also within the last 3 months):
     * Fasting plasma glucose > 130 mg/dL
     * 2-hour post-prandial or random blood glucose > 180 mg/dL
     * > 1 hypoglycemic event (blood glucose < 70 mg/dL) , or
  3. adults with T2D from the community who are new to insulin or being considered for insulin therapy by their healthcare provider.
  Interventions: Behavioral: Diabetes Pueblo

INTERVENTIONS:
Behavioral: Diabetes Pueblo — These adults will receive diabetes education, the Diabetes Pueblo Program, and will complete Curriculum (A), Diabetes Fundamentals, and Curriculum (B), Insulin Success.

SUMMARY:
Currently in the United States, the achieved level of glycemic control for adult Latinos with type 2 diabetes (T2D) is sub-optimal compared to the non-Latino Caucasian population. Among Latinos with T2D, there are unique barriers, such as socioeconomic and cultural factors, to starting and optimizing therapies, including insulin. Latinos have cultural beliefs and behaviors specific to this population that should be appropriately addressed in a diabetes self-management education and support program. Diabetes Pueblo is a diabetes education program that may be a solution to help address the barriers Latinos with T2D have to diabetes care and insulin use. The Diabetes Pueblo program consists of two targeted diabetes education curriculums for the local Latino community: (a) Diabetes Fundamentals and (b) Insulin Success, a culturally appropriate program course addressing barriers to initiating and optimizing insulin and T2D therapies. We will explore if Diabetes Pueblo Program improves knowledge of lifestyle advice for healthy eating and physical activity, increase the propensity to use insulin when clinically indicated, and improve success rates with insulin therapy by addressing common fears and negative perceptions of T2D therapies in this population.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a group of chronic disorders typified by raised blood glucose levels. An estimated 30 million people in the United States (US) (9.4% of the population) have diabetes. Type 1 diabetes (T1D) is defined by a rapid onset, often in childhood, and insulin dependence; while type 2 diabetes (T2D) is considered to have a slow onset and insulin insensitivity. Insulin is a required form of treatment for all T1D, and T2D patients who cannot achieve glycemic control through exercise and diet or other medications alone. Currently in the United States, the achieved level of glycemic control for adult Latinos with type 2 diabetes (T2D) is sub-optimal compared to the non-Latino Caucasian population. Among Latinos with T2D, there are unique barriers to starting and optimizing therapies, including insulin. Barriers include socioeconomic and cultural factors, as well as inadequate encouragement from health care providers. There are also challenges associated with access to timely and appropriate diabetes education. Some of these barriers may improve by using trained community health workers from the Latino community, as there is evidence that they are effective in supporting adherence and persistence with therapies (including insulin) and in encouraging lifestyle changes for T2D patients within their own communities.

The 2017 National Standards of Care for Diabetes Self-Management Education and Support (DSME/S) outline quality, evidenced based guidelines for DSME/S programs and guide those who will be providing these services. Benefits of DSME/S programs include improved clinical outcomes such as HbA1c and quality of life while reducing hospitalizations and health care costs. Hispanics are known to have a higher prevalence of diabetes, but use of DSME/S programs are vastly underutilized which means that many individuals in the Latino community with T2D are likely not receiving critical DSME/S services. It is crucial that DSME/S services be aligned with the needs of the target population in order to increase adherence and improve health outcomes. Latinos have cultural beliefs and behaviors specific to this population that should be appropriately addressed in a DSME/S program.

Diabetes Pueblo is a diabetes education program that may be a solution to help address the barriers Latinos with T2D have to diabetes care and insulin use. The Diabetes Pueblo program consists of two targeted diabetes education curriculums for the local Latino community: (a) Diabetes Fundamentals and (b) Insulin Success, a culturally appropriate program course addressing barriers to initiating and optimizing insulin and T2D therapies. Trained community health workers, also known as promotores, will deliver both programs. Ultimately, we will explore if Diabetes Pueblo Program improves knowledge of lifestyle advice for healthy eating and physical activity, increase the propensity to use insulin when clinically indicated, and improve success rates with insulin therapy by addressing common fears and negative perceptions of T2D therapies in this population.

This is a prospective pilot study. The Diabetes Pueblo program applied in this study is one program that consists of two newly created, targeted education curriculums for T2D Latino adults delivered over the course of 11 weeks by designated promotores, community health workers, to approximately 20 study participants at Sansum Diabetes Research Institute.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals > 18 years of age
2. Self-reported Latino heritage
3. Fluent in Spanish
4. Type 2 diabetes diagnosis
5. Available to attend the educational series and all study visits
6. Willingness to have height, weight, waist circumference, and HbA1c measured before and after the educational course
7. Individuals with poor glycemic control, as defined by the following:

   * HbA1c ≥ 8% at or prior to enrollment assessment (most recent lab within 3 months or provided at Sansum Diabetes Research Institute (SDRI) screening visit),

   OR
   * HbA1c < 8% (within the last 3 months), AND with at least one of the following (also within the last 3 months):

     * Fasting plasma glucose ≥ 130 mg/dL
     * 2-hour post-prandial or random blood glucose ≥ 180 mg/dL
     * ≥1 hypoglycemic event (blood glucose < 70 mg/dL)

   OR
   * Individuals new to insulin or being considered for insulin therapy by their healthcare provider
8. Willing and able to provide consent to take part in the study
9. Based on the research staff's judgment, participant must have a good understanding, ability, and willingness to adhere to the protocol

Exclusion Criteria:

1. Has a cognitive impairment, hearing difficulty, visual impairment, acute psychopathology, medical condition, or insufficient knowledge of the education program language that, in the opinion of the screener, would interfere with the ability to provide consent and participate/complete the program
2. Participation in other studies involving medications or device within 3 months prior to Visit 1
3. Known or suspected abuse of alcohol, narcotics, or illicit drugs
4. Current use of insulin pump
5. For females: Pregnancy or positive pregnancy test
6. Pharmaceutical employees or those employed in a position where they have a direct role in treating participants with diabetes.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Success (evaluated by a Yes/No format) recruiting and completing a new targeted diabetes and insulin education program, Diabetes Pueblo, for Latino adults with type 2 diabetes. | 11 weeks
  The Diabetes Pueblo program consists of two newly created, targeted education curriculums, Diabetes Fundamentals and Insulin Success, for Latino adults with type 2 diabetes. It will be delivered over the course of 11 weeks by designated promotores, community health workers, to approximately 20 study participants at Sansum Diabetes Research Institute.

SECONDARY OUTCOMES:
Diabetes self management evaluated by questionnaire | Visit 1, week 0 Screening; Visit 2, week 8 End of Diabetes Fundamentals class
  The Diabetes Self-Management Questionnaire consists of 16 questions to evaluate diabetes self-care including glucose management, dietary control, physical activity, and health-care use. Questions are rated on a 4 point scale - 0 Does not apply to me, 1 Applies to me to some degree, 2 Applies to me to a considerable degree, 3 Applies to me very much. This yields an overall rating of self-care with higher scores indicating more effective diabetes self-care.
Insulin treatment evaluated by questionnaire | Visit 1, week 0 Screening; Visit 2, week 8 End of Diabetes Fundamentals class; Visit 3, week 11 End of Insulin Success class
  The Insulin Treatment Appraisal Scale is a validated 20-item questionnaire that will be used in insulin naïve and insulin-treated patients with type 2 diabetes to assess positive and negative perceptions regarding insulin treatment. Items are rated on a 5-point scale ("strongly disagree" to "strongly agree") and the mean of individual item scores is calculated to obtain a total score, with lower scores indicating less negative perceptions regarding insulin treatment.
Participant evaluation of Diabetes Pueblo evaluated by questionnaire | Class 4, week 4; Class 8, week 8; Class 10, week 10
  The first questionnaire includes curriculum content questions which are specific to courses 1-4, 5-8, and 9-10.
Participant evaluation of Diabetes Pueblo evaluated by questionnaire | Class 11, week 11
  The second questionnaire assesses overall program feedback on the entire program.

OTHER OUTCOMES:
Fingerstick for evaluation of HbA1c related to diabetes | Visit 1, week 0 Screening; Visit 2, week 8 End of Diabetes Fundamentals class; Visit 3, week 11 End of Insulin Success class
  HbA1c % will measured in a capillary fingerstick blood sample
Height measured by Physical exam | Visit 1, week 0 Screening; Visit 2, week 8 End of Diabetes Fundamentals class; Visit 3, week 11 End of Insulin Success class
  Height measured in centimeters or inches by physical exam
Weight measured by Physical exam | Visit 1, week 0 Screening; Visit 2, week 8 End of Diabetes Fundamentals class; Visit 3, week 11 End of Insulin Success class
  Weight measured in kilograms or pounds by physical exam
Waist circumference measured by Physical exam | Visit 1, week 0 Screening; Visit 2, week 8 End of Diabetes Fundamentals class; Visit 3, week 11 End of Insulin Success class
  Waist circumference measured in centimeters or inches by physical exam
Socio-demographics assessed by questionnaire | Visit 1, week 0 Screening
  Socio-demographics measured by questionnaire - including age, gender, self-identified race/ethnicity, contact information, education, occupation, preferred language, insurance status, influenza & pneumonia immunization status, alcohol & tobacco use, birth place, physical activity, food security, and mobile phone use.
Foot examination evaluated by Questions | Visit 1, week 0 Screening
  Foot examination with 'yes or no' and frequency questions
Neuropathy Questions | Visit 1, week 0 Screening
  Questions about neuropathy
Retinopathy Questions | Visit 1, week 0 Screening
  Questions about retinopathy and eye exams
Nephropathy Questions | Visit 1, week 0 Screening
  Questions about nephropathy
Medical history and medication status and history assessed by questionnaire | Visit 1, week 0 Screening
  Medical history, including date of diabetes diagnosis, type of diabetes, diabetes education, diabetes self-care, depression and stress, falls, physician visits, hospital and emergency room visits, and current medications verified by visual inspection and medication history assessed by interview questionnaire
Menopausal status, pregnancy status, and gestational diabetes history for women determined by questionnaire | Visit 1, week 0 Screening
  Menopausal status, pregnancy status (number of live births, number of stillbirths, birthweights of live births, and any diagnosis of type 1 diabetes), and gestational diabetes history for female participants will be determined by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Creason, RD, Principal Investigator — Sansum Diabetes Research Institute
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No